CLINICAL TRIAL: NCT02404948
Title: Comparison of a Pulse Wave Based Approach for Detection of Coronary Artery Disease Compared to Standard Methods
Brief Title: PRV-based Detection of CAD in Comparison to Standard Methods
Acronym: PRV-KORO
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Marcus Doerr, Professor, University Medicine Greifswald
Other Study IDs: PRV-Koro-Study-001
Record Dates: First submitted 2015-03-23; First posted 2015-04-01 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; diagnosis; non-invasive
MeSH Terms: conditions — Coronary Artery Disease; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Diagnostic algorithm — Validation of a diagnostic algorithm used to detect coronary artery disease and/or myocardial ischemia based on pulse wave analyses.

SUMMARY:
This is a validation study comparing a pulse wave based algorithm for the detection of coronary artery disease with parameters from coronary angiography, echocardiography and cardiogoniometry.

DETAILED DESCRIPTION:
The study will validate a pulse wave based algorithm for the detection of coronary artery disease (CAD) with parameters from standard methods. Subjects will be patients admitted to coronary angiography due to suspected CAD. Pulse wave signals will be analyzed according to novelly established algorithm regarding the presence of CAD and/or myocardial ischemia. These results be compared to the diagnoses made by coronary angiography (primary endpoint): presence of minimum one coronary artery stenose >=50%. For secondary analyses, results will be compared to parameters form echocardiography and cardiogoniometry.

ELIGIBILITY:
Inclusion Criteria:

* Coronary angiography indication present
* informed written consent

Exclusion Criteria:

* Previous coronary angiography
* Known CAD (history of coronary angioplasty, stent implantation and/or bypass surgery)
* atrial fibrillation (at time of measurement)
* severe ventricular extrasystole (e.g. >=10% ventricular extrasystoles, bigemina)
* pregnancy, lactation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects referred to first coronary angiography due to suspected CAD
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Presence of CAD - angio (minimum 1 stenosis >=50%) | 1 day
  Presence of CAD in coronary angiography: minimum 1 stenosis >=50%

SECONDARY OUTCOMES:
Presence of CAD number - angio (Number of coronary vessels with at least 1 stenosis >=50% in coronary angiography) | 1 day
  Number of coronary vessels with at least 1 stenosis >=50% in coronary angiography
Wall motion abnormality - echo (Presence of wall motion abnormality in at least 1 segment (2D echocardiography) | 1 day
  Presence of wall motion abnormality in at least 1 segment (2D echocardiography)
Wall motion index - echo (Wall motion index (2D and 3D echocardiography) | 1 day
  Wall motion index (2D and 3D echocardiography)
Global longitudinal strain (2D and 3D echocardiography) | 1 day
  Global longitudinal strain (2D and 3D echocardiography)
Abnormal cardiogoniometry | 1 day
  Abnormal results of cardiogoniometry

CONTACTS AND LOCATIONS:
Locations (1):
- Marcus Dörr, Greifswald, Germany